CLINICAL TRIAL: NCT04506125
Title: Liberal Versus Restrictive Transfusion Threshold in High-risk Oncologic surgerY: a Multicenter, Randomized, Controlled, Pilot Study
Brief Title: Liberal Versus Restrictive Transfusion Threshold in Oncologic surgerY
Acronym: LIBERTY1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC20.0086
Record Dates: First submitted 2020-07-29; First posted 2020-08-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Oncologic Complications; Anemia
Keywords: Transfusion; Pilot study; critically ill patients; oncologic surgery
MeSH Terms: conditions — Anemia | interventions — Hemoglobins

STUDY DESIGN:
Intervention Model Description: Pilot, multicentre, randomized, controlled, single-blind, pilot study comparing two strategies for transfusion of red blood cell concentrates
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Group (Experimental): transfusion of an erythrocyte concentrate in case of haemoglobin below 9.5 g/dL
  Interventions: Other: Haemoglobin 9.5 g/dL
- Restrictive group (Active Comparator): transfusion of an erythrocyte concentrate in case of haemoglobin below 7.5 g/dL
  Interventions: Other: Haemoglobine 7.5g/dL

INTERVENTIONS:
Other: Haemoglobin 9.5 g/dL — transfusion of red blood cell concentrate if the haemoglobin level is less than 9,5 g/dL
  Arms: Liberal Group
Other: Haemoglobine 7.5g/dL — transfusion of red blood cell concentrate if the haemoglobin level is less than 7,5 g/dL
  Arms: Restrictive group

SUMMARY:
Anemia is common in oncology. Up to three-quarters of cancer patients are exposed to an episode of anemia. In oncology surgery, perioperative bleeding is a major risk factor for anemia. Indeed, 13 to 40% of patients are transfused in perioperative oncologic surgery.

There is an association between anemia and prognosis. Several epidemiological studies have shown a strong association between anemia and altered quality of life. In oncology cohort studies, anemic patients had a significantly lower quality of life compared to patients without anemia. In non-cardiac surgery, preoperative anaemia was significantly associated with post-operative mortality. There is also an association between preoperative anaemia and the occurrence of post-operative complications. In oncology surgery, cohort studies conducted in colorectal surgery and neurosurgery found an association between the occurrence of perioperative anemia and post-operative morbidity and mortality.

The optimal transfusion strategy is unknown in oncology patients. Several multicentre randomised trials, conducted in resuscitation patients or in perioperative settings, have compared a "restrictive" to a "liberal" transfusion strategy. These studies did not show a superiority of one strategy over another on patient outcomes but a lower exposure to red blood cell concentrates in patients transfused with the restrictive transfusion strategy. Thus, the French High Authority for Health (HAS) has adopted a haemoglobin level of 7 g/dl as the transfusion threshold for any transfusion of red blood cell concentrate carried out in the operating theatre and in intensive care in the absence of special cases such as the presence of acute coronary syndrome. For oncology patients, no recommendation could be made due to the lack of evidence-based literature and the optimal transfusion strategy for these patients remains unknown. Only 2 monocentric trials performed in oncology (critical care and perioperative) suggest a benefit of a liberal strategy (transfusion for a haemoglobin level < 9 g/dl) on the short-term vital prognosis, but these studies suffer from numerous limitations leaving the question unresolved.

Before conducting a large phase III trial, a pilot study is needed to validate the methodology of this multicentre clinical trial and to assess its feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Anticipated or proven admission to immediate postoperative resuscitation after scheduled or emergency oncology surgery, for the removal of a neoplastic lesion among the following surgical procedures:

  * Visceral surgery: Hepatectomy, duodenopancreatectomy, gastrectomy, esophagectomy, colectomy
  * Urological surgery: Radical prostatectomy, cystectomy, nephrectomy.
  * Gynaecological surgery: Ovariectomy, hysterectomy, mastectomy, pelvectomy
  * Thoracic surgery: Pneumonectomy, lobectomy
  * ENT Surgery: Total laryngectomy, pharyngectomy, glossectomy
  * Spinal surgery: corporectomy wherever it is performed.
* Hemoglobin level < 9.5 g/dl between the day before surgery (D-1) and discharge from resuscitation at no more than 30 days postoperatively

Exclusion Criteria:

* - Myocardial infarction and/or unstable angina in the 4 weeks prior to surgery
* Refusal to participate in the study
* Minor patient (age < 18 years)
* Refusal to transfuse red blood cell concentrates (Jehovah's Witness)
* Pregnant or breastfeeding women
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Methodology of the pilot study | up to 30 days
  The difference in mean hemoglobin levels during the perioperative period up to 30 days postoperatively between the two groups will be assessed

SECONDARY OUTCOMES:
Epidemiological data of the pilot study | up to 90 days
  The percentage of patients with oncologic surgery admitted to intensive care unit requiring transfusion of red blood cell concentrates eerioperatively among aatients with oncologic surgery admitted to intensive care unit will be assessed
Epidemiological data of the pilot study | up to 90 days
  Percentage of eligible patients included in the study will be assessed
Epidemiological data of the pilot study | up to 90 days
  Delay between surgery and randomization will be assessed
Epidemiological data of the pilot study | up to 90 days
  Percentage of protocol violations in each group will be assessed
Epidemiological data of the pilot study | up to 90 days
  Average number of erythrocyte concentrates delivered to each group intraoperatively, in intensive care and during hospitalization will be assessed
Epidemiological data of the pilot study | up to 90 days
  Post-operative complications, occurring between surgery and the 30th day after surgery or before discharge from hospital will be assessed
Adverse Reaction Monitoring | up to 30 days
  To compare the occurrence of transfusion-related adverse events in each group
Evaluation of the functional status | up to 30 days
  Test functional status assessment at 30 days postoperatively using the World Health Organization Disability Assessment Schedule (WHODAS) questionnaire.
  This questionnaire asks about difficulties due to health/mental health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long lasting, injuries, mental or emotional problems, and problems with alcohol or drugs. The patient must think back over the past 30 days and answer the questions thinking about how much difficulty you had doing the following activities.
Evaluation of the functional status after surgery ans anesthesia | up to 30 days
  Test functional status assessment at 30 days postoperatively using the Quality of recovery questionnaire.
  The Quality of Recovery-15 (QoR-15) is a psychometrically tested and validated questionnaire.
  The QoR-15 was psychometrically evaluated using data collected from patients who responded at all four time intervals.This included: Acceptability and Feasibility; Validity; Reliability; Responsiveness
Monitoring of the quality of the study's execution | up to 30 days
  Compare the percentage of protocol violations in the 2 groups

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU d'Angers, Angers
  - CHRU de Brest, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836